CLINICAL TRIAL: NCT05360446
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase IIIb Study Evaluating the Effect of Inclisiran on Atherosclerotic Plaque Progression Assessed by Coronary Computed Tomography Angiography (CCTA) in Participants With a Diagnosis of Non-obstructive Coronary Artery Disease Without Previous Cardiovascular Events (VICTORION-PLAQUE)
Brief Title: Coronary Computed Tomography Study to Assess the Effect of Inclisiran in Addition to Maximally Tolerated Statin Therapy on Atherosclerotic Plaque Progression in Participants With a Diagnosis of Non-obstructive Coronary Artery Disease Without Previous Cardiovascular Events
Acronym: V-PLAQUE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CKJX839D12303; 2021-004601-47 (EudraCT Number)
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Inclisiran; KJX839; Atherosclerotic plaques; CCTA; CT-adapted Leaman score; LDL-C; FFRct; NOCAD; PCSK9 inhibitor; TAV
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sponsor personnel participating in the study conducted will be blinded also.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Drug: Placebo
- Inclisiran sodium (Experimental): Subcutaneous injection
  Interventions: Drug: Inclisiran sodium 300 mg

INTERVENTIONS:
Drug: Inclisiran sodium 300 mg — Subcutaneously administered on Days 1, Month 3 (Day 90), and every 6 months thereafter.
  Arms: Inclisiran sodium
Drug: Placebo — Subcutaneously administered on Day 1, Month 3 (Day 90), and every 6 months thereafter.
  Arms: Placebo

SUMMARY:
CKJX839D12303 is a research study to determine if the study treatment, called inclisiran, in comparison to placebo taken in addition to statin medication can effectively reduce the total amount of plaque formed in the heart's vessels as measured by coronary computed tomography angiography (CCTA) from baseline to month 24. This study is being conducted in eligible participants with a diagnosis of non-obstructive coronary artery disease (NOCAD), where the coronary arteries are blocked less than 50%, and with no previous cardiovascular events.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of inclisiran compared to placebo on top of maximally tolerated dose of statin therapy in reducing total coronary atheroma volume assessed by CCTA in participants with a diagnosis of Non-Obstructive Coronary Artery Disease (NOCAD) without previous cardiovascular events, who have an LDL-C ≥55 mg/dL (1.4 mmol//L), no significant pressure drop in Fractional Flow Reserve Computed Tomography (FFRCT) and a CT-adapted Leaman score >5 despite the use of maximally tolerated statin therapy(and if applicable, another LLT on top of statin therapy for at least 30 days in up to 20% of randomized participants).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years or ≤80 years of age at signing of informed consent.
* Fasting LDL-C local lab value at the Screening Visit of either i) ≥100 mg/dL (2.6 mmol/L) if on statin therapy but not on a maximally tolerated statin therapy; ii) ≥150 mg/dL (3.9mmol/L) if statin naive and without documented statin intolerance; or iii) ≥55 mg/dL (1.4 mmol/L) if on a stable (≥4 weeks) dose of maximally tolerated statin therapy or if statin intolerant.
* Fasting LDL-C local lab value ≥55 mg/dL (1.4 mmol/L) at the assessment performed during the Statin Optimization Period 3 Visit for participants going through the Statin Optimization Period.
* Participants having NOCAD without previous cardiovascular events: NOCAD is defined as:.

  1. Participant with CT-adapted Leaman score >5. and a diameter stenosis <50% or
  2. Participants with a CT-adapted Leaman score >5, a diameter stenosis ≥50% but with FFRCT ≥0.76.
* A standard of care CCTA may serve as the study baseline CCTA scan if it is performed within 3 months prior to the participant's Screening Visit and meets the inclusion criteria of FFRct >0.8 and CT-adapted Leaman score >5, which will be assessed by the Imaging Core Lab.
* At the Baseline Visit, participants must be on a stable (≥4 weeks) dose of maximally tolerated statin therapy. Participants not on maximally tolerated statin therapy and who do not have documented statin intolerance can be screened but must enter the study via a Statin Optimization Period.
* Fasting LDL-C lab value ≥55 mg/dL (1.4 mmol/L) at the Baseline Visit, measured at the central laboratory. If the Baseline and Screening Visits occur on the same day, then the LDL-C assessment will be assessed on the central laboratory sample. If a participant qualifies at Screening but the fasting central lab LDL-C value at the Baseline visit does not meet eligibility, then eligibility will be determined based on the central lab result.
* Fasting triglycerides value <400 mg/dL (4.52 mmol/L) based on the local lab results at the Screening visit and on the central lab results at the CCTA visit.

Exclusion Criteria:

* Previous cardiovascular events history including myocardial infarction (MI), or prior coronary revascularization [percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)].
* Planned revascularization (PCI) or (CABG).
* Previous cerebrovascular events including:

  * Prior ischemic stroke thought not to be caused by atrial fibrillation, valvular heart disease or mural thrombus.
  * History of prior percutaneous or surgical carotid artery revascularization.
* History of Peripheral Artery Disease (PAD):

  * Prior documentation of a resting ankle-brachial index <0.85.
  * History of prior percutaneous or surgical revascularization of an iliac, femoral, or popliteal artery.
  * Prior non-traumatic amputation of a lower extremity due to peripheral artery disease.
* Cardiac disorders, including any of the following:

  * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, atrial fibrillation) within 3 months prior to randomization that is not controlled by medication or via ablation at the time of the Screening Visit.
  * Complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third-degree AV block) prior to randomization.
* Contraindication for CCTA (e.g., allergic reactions to the contrast dye) or CCTA not meeting entry standards after two attempts during the Baseline CCTA Visit as assessed by the Imaging Core Lab.
* Pacemaker or implantable cardioverter-defibrillator (ICD) in situ.
* Systolic Left Ventricle Ejection Fraction <30% at the Screening Visit.
* Uncontrolled severe hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to randomization (assessed at the Screening Visit) despite antihypertensive therapy.
* Heart failure New York Heart Association (NYHA) class III or class IV at the Screening Visit.
* Renal insufficiency (eGFR <30 mL/min/1.73m2) as measured by the Modification of Diet in Renal Disease (MDRD) formula at the Screening Visit and at the Statin Optimization 3 Visit.
* Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver at the Screening Visit.
* Local creatine kinase (CK) values of either, unless a more stringent threshold is mandated by a local regulatory authority
* Local CK values ≥5x ULN at the Statin Optimization 3 Visit unless a more stringent threshold is mandated by a local regulatory authority
* Participant with myopathy at the Statin Optimization 3 Visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Percentage change in total coronary atheroma volume | From baseline to month 24
  Evaluating inclisiran compared to placebo both on top of maximally tolerated statin therapy in reducing total coronary atheroma volume assessed by coronary computed tomography angiography (CCTA) in participants with a diagnosis of non-obstructive coronary artery disease (NOCAD) without previous cardiovascular events.

SECONDARY OUTCOMES:
Percentage change in LDL-C | From baseline to month 24
  Full fasting lipid panel will be collected throughout the study beginning at baseline.
Percentage change in low attenuation plaque volume evaluated by CCTA | From baseline to month 24
  Evaluating inclisiran compared to placebo in percentage change in low attenuation plaque volume evaluated by CCTA.
Percentage of participants with progression, regression, or no change of total plaque atheroma volume | From baseline to month 24
  Evaluating inclisiran compared to placebo in percentage of participants experiencing progression, regression, or no change of total atheroma volume.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (84):
- United States (27):
  - Heart Center Research Llc, Huntsville, Alabama
  - Alaska Heart and Vascular, Anchorage, Alaska
  - Cardiovascular Res Found, Beverly Hills, California
  - UC San Diego Health, La Jolla, California
  - Stanford Health Care, Stanford, California
  - Lundquist Inst BioMed at Harbor, Torrance, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - George Washington Univ Medical Ctr, Washington D.C., District of Columbia
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Reid Physician Associates, Richmond, Indiana
  - Midwest Heart and Vascular Spec, Overland Park, Kansas
  - Anderson Medical Research, Ft. Washington, Maryland
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - R Ins For Heart And Vascular Health, Reno, Nevada
  - Cardio Metabolic Institute, Somerset, New Jersey
  - Icahn School of Med at Mt Sinai, New York, New York
  - State Uni of NY at Stony Brook, Stony Brook, New York
  - Westchester Medical Center, Valhalla, New York
  - Aultman Hospital, Canton, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Orion Medical, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Swedish Medical Center-Cardiovascular Research, Seattle, Washington
  - Univ of Washington Medical Center, Seattle, Washington
- Argentina (2):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (4):
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Chemside, Queensland
  - Novartis Investigative Site, Milton, Queensland
  - Novartis Investigative Site, Leabrook, South Australia
- Belgium (5):
  - Novartis Investigative Site, Turnhout, Antwerpen
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Hasselt, Limburg
  - Novartis Investigative Site, Yvoir, Namur
  - Novartis Investigative Site, Aalst, Oost Vlaanderen
- Brazil (3):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo
- Canada (3):
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Santiago, Santiago Metropolitan, Chile
- China (4):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- France (4):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Toulouse
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- India (7):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, New Delhi
- Ireland (2):
  - Novartis Investigative Site, Dublin, Ireland
  - Novartis Investigative Site, Galway
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Torino, TO
- Japan (4):
  - Novartis Investigative Site, Miyhazaki, Miyazaki
  - Novartis Investigative Site, Urasoe, Okinawa
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Kyoto
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (6):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Valencia
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lugano
- United Kingdom (2):
  - Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear
  - Novartis Investigative Site, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Revaiah PC, Serruys PW, Onuma Y, Andreini D, Budoff MJ, Sharif F, Chernofsky A, Vikarunnessa S, Wiethoff AJ, Yates D, Achouba A. Design and rationale of a randomized clinical trial assessing the effect of inclisiran on atherosclerotic plaque in individuals without previous cardiovascular event and without flow- limiting lesions identified in an in-hospital screening: The VICTORION-PLAQUE primary prevention trial. Am Heart J. 2026 Jan;291:199-212. doi: 10.1016/j.ahj.2025.08.001. Epub 2025 Aug 30. PMID 40769373